CLINICAL TRIAL: NCT04918056
Title: Screening and Identification of Genetic Modifiers Which Affecting the Phenotype Severity of Beta Thalassemia Patients
Brief Title: Genetic Variants Affecting the Clinical Severity of Beta Thalassemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: 303rd Hospital of the People's Liberation Army (Other); Liuzhou Municipal Maternity and Child Healthcare Hospital (Unknown); Zhuhai Municipal Maternal and Child Healthcare Hospital (Unknown); Dong Guan Maternal and Child Health Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: PDD-Beta thalassemia
Record Dates: First submitted 2021-06-03; First posted 2021-06-08 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Beta Thalassemia
Keywords: beta thalassemia; Hb F; Onset age; Genetic Modifier
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- beta thalassemia patients
  Interventions: Diagnostic Test: Hematological Analysis and Genetical Analysis

INTERVENTIONS:
Diagnostic Test: Hematological Analysis and Genetical Analysis — Hematological Analysis: Hematological parameters were determined with an automated hematology analyzer (Sysmex, Japan), and hemoglobin analysis was performed with either high-performance liquid chromatography (Bio-Rad, USA) or capillary electrophoresis (Sebia, France and Helena, USA).
  Genetical Analysis: Genomic DNA was extracted from peripheral blood (PB) by using a standard phenol/chloroform method. The genotypes of samples are analyzed by NGS assay.

SUMMARY:
β-thalassemia is one of the most common single gene disorder in Southern China. The phenotypic severity of beta thalassemia widely varies from mild to severe forms. Patients with the same beta thalassemia genotype show wide phenotypic variability that ranges from moderate to severe disease due to various genetic modifiers of disease severity. The aim of this study is to looking for the genetic factors which could affect the severity of beta thalassemia.

DETAILED DESCRIPTION:
The understanding of the genotype-phenotype correlation is a very important issue to the precise diagnosis of beta thalassemia. However, the genotype-phenotype correlation of Beta thalassemia is so complex that the pathogenesis of some patients remains uncertain and cannot be explained by known mechanisms. The study of the role of the genetic variants in modulating beta thalassemia phenotype could brought us considerable novel and interesting information in this area. We will collecting more than 1000 beta thalassemia patients , analyzing their clinical data and genome data, and association study will be conducted to screen the positive genetic variants which exert a significant effect on both the HbF levels and onset ages of beta thalassemia patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with β-thalassemia

Exclusion Criteria:

* Iron Deficiency Anemia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: beta thalassemia patients from Southern China.
Sampling Method: Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-01-11 (Estimated); Study Completion 2023-06-25 (Estimated)

PRIMARY OUTCOMES:
Genetic variants which could influence the phenotype of beta thalassemia | 1 year
  Identified a group of single-nucleotide polymorphisms (SNPs) that contribute to β-thalassemia

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Medical University, Guangzhou, Guangdong, China